CLINICAL TRIAL: NCT07009002
Title: A Phase I/II Single-center Study Evaluating the Safety and Efficacy of BCOR and ZC3H12 Genes Knock-out CD19-targeting CAR-T Cell Therapy in Adults With Refractory/Relapsed Refractory/Relapsed B-cell Lymphoma
Brief Title: BCOR and ZC3H12 Genes Knock-out CD19-targeting CAR-T Cell Therapy in r/r B Cell Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Director of Biotherapeutic Department, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-092
Record Dates: First submitted 2025-05-21; First posted 2025-06-06 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: B Cell Lymphoma
Keywords: CAR-T cells; CD19
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — fludarabine; fludarabine phosphate; Injections; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR19TIF cells (Experimental): Patients with r/r B Cell Lymphoma conditioning chemotherapy regimen of fludarabine and cyclophosphamide will be administered followed by investigational treatment, CAR19TIF cells.
  Interventions: Biological: CAR19TIF cells; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: CAR19TIF cells — Phase 1 dose escalation/decline (3+3) : starting dose:
  5×10^5 cells/kg, According to effective expansion and clinical efficacy data, a descending dose escalation model will be adopted: such as 1×10^5 cells/kg, 5×10^4 cells/kg. If the 5×10^5 cells/kg dose group does not achieve efficient expansion and clinical benefit, an ascending dose escalation model will be adopted, such as 2×10^6 cells/kg, 6×10^6 cells/kg. Phase 2 : dose of RP2D.
  Other Names: BCOR and ZC3H12 genes knock-out CD19 CAR T cells
Drug: Fludarabine — Intravenous fludarabine 25~30 mg/m^2/day on days
  -5, -4, and -3.
  Other Names: Fludarabine Phosphate for Injection
Drug: Cyclophosphamide — Intravenous cyclophosphamide 250~500 mg/m^2/day on days -5, -4, and -3.
  Other Names: Cyclophosphamide for Injection

SUMMARY:
In this single-center, single-arm, prospective, Phase 1/2 study, the safety and efficacy of autologous BCOR and ZC3H12 genes knock-out CD19-targeting chimeric antigen receptor (CAR) T-cell therapy will be evaluated in patients with refractory/relapsed (r/r) B-cell Lymphoma. For simplicity, we have termed these CD19 CAR T cells lacking ZC3H12A and BCOR as CAR19TIF( immortal-like and functional CD19 CAR T ) cells, reflecting their immortal-like and functional characteristics.

In phase 1, 3 eligible patients will be enrolled and receive CAR19TIF cells at a initial dose of 5×10^5 cells/kg. Based on the results, subsequently an additional 3-15 patients will be enrolled in a "3+3" dose-escalation/decline design to adjust the dose of CAR19TIF cells to achieve optimal safety and efficacy. The recommended Phase 2 dose (RP2D) will then be established. 10 to 12 subjects will be enrolled and receive CAR19TIF cells infusion at dose of RP2D.

DETAILED DESCRIPTION:
Phase 1 (dose escalation/decline)

In phase 1, 6-18 subjects will be enrolled. Referring to the starting dose of most CAR-T cell therapies, and to avoid exposing patients to the risk of "ineffective expansion dose", 3 patients will receive CAR19TIF cells therapy at a starting dose of 5×10^5 cells/kg.According to the copy number of CAR-T cells were assessed by number in peripheral blood and clinical efficacy data, additional 3-15 patients will be enrolled in a "3+3" dose-escalation/decline design to adjust the dose of CAR19TIF cells to achieve optimal safety and efficacy :

After obtaining effective expansion data and clinical efficacy data, a descending dose escalation model will be adopted: such as 1×10^5 cells/kg, 5×10^4 cells/kg. If the 5×10^5 cells/kg dose group does not achieve efficient expansion and clinical benefit, an ascending dose escalation model will be adopted, such as 2×10^6 cells/kg, 6×10^6 cells/kg.

3 subjects are enrolled in a cohort corresponding to a dose level. If 1 subject in a cohort of 3 subjects experiences a DLT, 3 additional subjects will be enrolled at the current dose level.

For safety purposes, the administration of CAR19TIF cells will be staggered by 28 days between the first two subjects in each cohort. And for each of the remaining cohorts, the administration of CAR19TIF cells will be staggered by 28 day.

Phase 2 (expansion cohort) In phase 2, 10 to 12 subjects will be enrolled and receive cell infusion at dose of RP2D, which will be determined based on the maximum tolerated dose (MTD), occurrence of DLT, the obtained efficacy results, pharmacokinetics/pharmacodynamics and other data according to the phase 1.

Objectives The primary objectives of the phase 1 were to evaluate the tolerability and safety of CAR19TIF cells in patients with r/r B-cell Lymphoma

, and determine RP2D. The primary purpose of the phase 2 study was to evaluate the efficacy of CAR19TIF cells in the above population.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 (inclusive).
2. Subjects who meet the following requirements:

   2.1 Histologically confirmed refractory/relapsed B cell Non-Hodgkin's lymphomas (NHL), including the following types defined by World Health Organization (WHO) 2016:
   * Diffuse large B-cell lymphoma not otherwise specified (DLBCL NOS);
   * Primary mediastinal (thymic) large B-cell lymphoma (PMBCL);
   * Transformed follicular lymphoma (TFL);
   * High-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements (HGBCL);
   * Follicular lymphoma (FL);
   * Mantle cell lymphoma (MCL) (pathologically confirmed, with documentation of monoclonal B cells that have a chromosome translocation t(11;14)(q13;q32) and/or overexpress cyclin D1);
   * Marginal zone lymphoma (MZL), including nodal or splenic marginal zone B-cell lymphoma and mucosa-associated lymphoid tissue (MALT) lymphoma.

   2.2 Relapsed disease is defined as disease progression (PD) after achieving disease remission (including CR and PR) with the latest standard regimen.

   2.3 Refractory disease is defined as no CR to first-line therapy: Evaluation of PD (never reached response or SD) after standard first-line treatment, or
   * SD as best response after at least 4 cycles of first-line therapy (eg,4 cycles of R-CHOP), or
   * PR as best response after at least 6 cycles and biopsy-proven residual disease or disease progression ≤ 6 months of therapy, or
   * Refractory post-autologous stem cell transplant (ASCT): i. Disease progression or relapsed less than or equal to 12 months of ASCT (must have biopsy proven recurrence in relapsed individuals); ii. If salvage therapy is given post-ASCT, the individual must have had no response to or relapsed after the last line of therapy.

   2.4 Individuals who are intolerant to standard treatment can also be included in the study in the investigator's judgment.
3. Individuals must have received adequate prior therapy:

   3.1 For MCL, prior therapy must have included:
   * Anthracycline or bendamustine-containing chemotherapy and
   * Anti-CD20 monoclonal antibody (unless investigator determines that tumor is CD20-negative) and
   * Bruton's tyrosine kinase inhibitor (BTKi). 3.2 For other types, prior therapy must have included:
   * Anti-CD20 monoclonal antibody (unless investigator determines that tumor is CD20-negative) and
   * Anthracycline containing chemotherapy regimen. 3.3 For individual with transformed FL must have relapse or refractory disease after transformation to DLBCL.
4. At least 1 measurable lesion: lymph node site with a long axis >1.5cm, extranodal site with a long axis >1.0cm (according to the Lugano2014 criteria). Lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy.
5. CD19 positive (detected by immunohistochemistry [IHC]).
6. Toxicities due to prior therapy must be stable and recovered to ≤ Grade 1 (except for hematological toxicities and clinically non-significant toxicities such as alopecia).
7. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
8. Absolute neutrophil count (ANC) ≥ 1 x 10^9/L, Platelet count ≥50 x 10^9/ L, hemoglobin (Hgb) ≥ 80g/L (hemocytopenia caused by lymphoma invasion of bone marrow is not subject to conditions above).
9. Adequate renal, hepatic, pulmonary and cardiac function defined as:

   9.1 Serum creatinine≤1.5 upper limit of normal (ULN) or creatinine clearance (as estimated by Cockcroft Gault) ≥ 60 mL/min.

   9.2 Serum alanine aminotransferase / aspartate aminotransferase (ALT/ AST) ≤ 3 upper limit of normal (ULN); Total bilirubin ≤ 1.5 ULN, except in subjects with 3) Gilbert's syndrome.

   9.3 Cardiac ejection fraction ≥ 50%, no evidence of pericardial effusion as determined by an echocardiogram (ECHO), and no clinically significant electrocardiogram (ECG) findings.

   9.4 Coagulation Function: International Normalized Ratio (INR) ≤ 1.5 times the upper limit of normal (ULN), and Activated Partial Thromboplastin Time (APTT) ≤ 1.5 times ULN.

   9.5 Baseline oxygen saturation >91% on room air.
10. Subjects of both genders who are willing to practice birth control from the time of consent through 6 months after the completion of conditioning chemotherapy. Females of childbearing potential must have a negative serum or urine pregnancy test (females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential).
11. Voluntarily participate in this clinical trial and sign an informed consent form.

Exclusion Criteria:

1. Expected survival time < 3 months per Principal Investigator's opinion.
2. History of malignancy other than nonmelanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast) or follicular lymphoma unless disease free for at least 3 years.
3. History of allogeneic hematopoietic stem cell transplantation, or organ transplantation.
4. Prior CD19 targeted therapy.
5. Patients who have used any of the following agents or treatments within a specific period of time:

   5.1 Received any chemotherapy drugs or small molecule targeted drugs within 2 weeks prior to lymphodepletion; 5.2 Received any monoclonal antibodies, antibody drug conjugates (ADCs), or bispecific antibodies within 3 weeks prior to lymphodepletion; 5.3 Received radiotherapy within 6 weeks prior to lymphodepletion. However, if disease progressed at the site of radiotherapy, or if there are positive lesions detected by PET-CT at non-radiotherapy sites, enrollment is allowed.
6. Prior CAR-T therapy or other genetically modified T cell therapy.
7. Subjects with detectable cerebrospinal fluid malignant cells, or brain metastases, or with a history of central nervous system (CNS) lymphoma or primary CNS lymphoma.
8. History of severe, immediate hypersensitivity reaction attributed to lymphodepletion drugs or any component of CAR19TIF cells.
9. Presence or suspicion of fungal, bacterial, viral, or other infection that is uncontrolled or requiring intravenous (IV) antimicrobials for management.
10. Uncontrolled or active infectious diseases, such as human immunodeficiency virus (HIV) infection, acute or chronic active hepatitis B or C, epstein-barr virus (EBV), and cytomegalovirus (CMV) infection.
11. History or presence of CNS disorder such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement.
12. Subjects with cardiac atrial or cardiac ventricular lymphoma involvement.
13. History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 12 months of enrollment.
14. Expected or possible requirement for urgent therapy within 6 weeks due to ongoing or impending oncologic emergency (eg, tumor mass effect, tumor lysis syndrome).
15. Primary immunodeficiency.
16. History of autoimmune disease (e.g. Crohn's, rheumatoid arthritis, systemic lupus) resulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years.
17. History of symptomatic deep vein thrombosis or pulmonary embolism requiring systemic anticoagulation within 6 months of enrollment.
18. Any medical condition likely to interfere with assessment of safety or efficacy of study treatment.
19. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
20. Vaccine ≤ 6 weeks prior to planned start of conditioning regimen.
21. In the investigator's judgment, the subject is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | 12 months
  AE is defined as any adverse medical event from the date of randomization to 12 months after CAR T cells infusion. Among them, cytokine release syndrome(CRS) and immune cell-associated neurotoxicity syndrome (ICANS) were graded according to American Society for Transplantation and Cellular Therapy (ASTCT) criteria. Other AEs were graded according to common terminology criteria for adverse events (CTCAE) v5.0.
Phase 1: Incidence of Incidence of DLT. | First infusion date of CAR-T cells up to 28 days.
  DLT is defined as any AE related to the investigational drug that occurs within 28 days after administration of the CAR19TIF cells and meets any one of the criteria listed in the DLT criteria:
  * Grade 3 CRS that does not resolve to grade 2 or lower within 2 weeks;
  * Grade 3 ICANS lasting for ≥ 7 days;
  * Any Grade ≥ 4 CRS or ICANS;
  * Any other Grade ≥ 4 and Grade 3 AEs related to the CAR19TIF cells that lasts for ≥ 14 days, except hematology toxicity.
RP2D | 12 months
  The recommended dose for phase 2 was determined through phase 1 study.
Phase 2: Complete response (CR) rate | 24 months
  CR is assessed by investigators and based on the Lugano 2014 assessment criterion. CR rate is defined as the proportion of patients who have achieved CR assessed by investigators.
Phase 2: Objective response rate (ORR) | 24 months
  ORR is defined as the proportion of patients who have achieved CR and partial response (PR) assessed by investigators.
Phase 2: Duration of Response (DOR) | 24 months
  DOR is defined as the date of their first CR or PR (which is subsequently confirmed) to PD assessed by investigators, or death regardless of cause.
Phase 2: Overall Survival (OS) | 24 months
  OS is defined as the time from CAR-T cells infusion to the date of death. Subjects who have not died by the analysis data cutoff date will be censored at the last contact date.
Phase 2: Progression Free Survival (PFS) | 24 months
  PFS is defined as the time from the CAR-T cells infusion date to the date of disease progression assessed by investigators, or death any cause. Participants not meeting the criteria for progression by the analysis data cutoff date were censored at the last evaluable disease assessment date.

SECONDARY OUTCOMES:
Phase 1 and phase 2: Pharmacokinetics:Level of CAR-positive T cells circulating in blood over time | 12 months
  Number (cells/ul)and copy number (copies/ug DNA) of CAR-T cells were assessed by number in peripheral blood. Blood samples were collected before and one year after cell infusion (until CAR-T cells were not detected for two consecutive times) to detect the number and copy number of CAR-T cells, and to evaluate the pharmacokinetics of CAR-T.
Phase 1 and phase 2: Pharmacodynamics:Level of CD19+ cells in peripheral blood | Up to 28 days after infusion.
  The level of CD19+ cells (%) in peripheral blood will be detected by flow cytometry.
Phase 1 and phase 2: Peak level of cytokines in serum (phase 1 and phase 2) | Up to 28 days after infusion
  The cytokines mainly include interleukin-2 (IL-2 ), IL-6, IL-8, IL-10, tumor necrosis factor-α (TNF-α), C reactive protein .
Phase 1: 3-month ORR | 3 months
  The definition of ORR has already been mentioned above
Phase 1: OS | 24 months
  The definition of OS has already been mentioned above
Phase 1: PFS | 24 months
  The definition of PFS has already been mentioned above
Phase 2: Incidence of AE | 24 months
  AE is defined as any adverse medical event from the date of enrollment to 24 months after CAR-T cells infusion.

OTHER OUTCOMES:
Relationship between infusion dose of CAR T cells and efficacy | 24 months
  Peripheral blood was collected at the day of infusion (day 1), day 4, day 7, day 11, day 14, day 28, at least once every month after 28 days, at least once every three months after half a year, and at least once every six months after a year. The researchers will analyze the relationship between the number of CAR T cells, copy number, cytokines level, and efficacy of CAR T cells. The number of CAR T cells was detected by flow cytometry, and the copy number was detected by quantitative PCR (qPCR).
To analyze the dynamic changes of CAR T cells after infusion | 24 months
  The dynamic changes of the number and copy number of CAR T cells in patients after CAR T treatment were analyzed. To summarize the characteristic of the peak(cells/ul) , expansion pattern, continuous expansion time (days )and evolution of CAR T cells in vivo.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Han, Ph.D, Principal Investigator — Biotherapeutic Department, Chinese PLA General Hospital
Locations (1):
- Biotherapeutic Department of Chinsese PLA Gereral Hospital, Beijing, Beijing Municipality, China